CLINICAL TRIAL: NCT01084395
Title: Reducing HIV Risk Among Mexican Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Antonia M. Villarruel, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H03-00001528-MI; R01NR008059 (NIH)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections; AIDS; Sexually Transmitted Diseases
Keywords: Parent; Adolescent; Mexico; Safer Sex Communication; Randomized Controlled Trial; HIV/AIDS; STD; Sexual Behavior
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Adolescent Safer Sex Intervention (Experimental)
  Interventions: Behavioral: Adolescent Safer Sex Intervention
- Parent Safer Sex Intervention (Experimental)
  Interventions: Behavioral: Parent Safer Sex Communication Intervention
- Adolescent Health Promotion Control (Other)
  Interventions: Other: Adolescent Health Promotion Control Condition
- Parent Health Promotion Control (Other)
  Interventions: Other: Parent Health Promotion Control Condition

INTERVENTIONS:
Behavioral: Adolescent Safer Sex Intervention — Adolescents are randomly assigned to the HIV risk-reduction intervention condition. Adolescents receive a theory-based intervention designed to reduce HIV risk-associated behavior. The intervention consists of six 50-minute modules implemented over the course of two days. The intervention is highly interactive and includes games, videos, discussion, and role-plays.
  Other Names: Cuidate
  Arms: Adolescent Safer Sex Intervention
Behavioral: Parent Safer Sex Communication Intervention — Parents are randomly assigned to the Safer Sex Communication Intervention. Parents learn about HIV and other consequences of unprotected sexual behavior. The intervention contains content that focuses on enhancing parent-adolescent communication.
  Arms: Parent Safer Sex Intervention
Other: Adolescent Health Promotion Control Condition — Adolescents are randomly assigned to the Health Promotion control condition. Adolescents receive an intervention aimed at significant health problems affecting Mexicans that are related, not to sexual behavior, but to other behaviors. These health problems include heart disease, certain cancers, and diabetes. Adolescents are taught that these health problems can be prevented by changing personal behaviors, primarily exercise, diet, cigarette smoking, and alcohol and drug use.
  Arms: Adolescent Health Promotion Control
Other: Parent Health Promotion Control Condition — Parents are randomly assigned to the Health Promotion control condition. Parents receive an intervention aimed at significant health problems affecting Mexicans that are related, not to sexual behavior, but to other behaviors. These health problems include heart disease, certain cancers, and diabetes. Parents will be taught that these health problems can be prevented by changing personal behaviors, primarily exercise, diet, cigarette smoking, and alcohol and drug use. The intervention also provides content that emphasizes the importance of families.
  Arms: Parent Health Promotion Control

SUMMARY:
The broad objective of this project is to test the efficacy of a theory-based HIV risk-reduction intervention, which includes both an adolescent component and parental component, designed to reduce the adolescents' risk of sexually transmitted HIV.

DETAILED DESCRIPTION:
Sexually transmitted HIV infection among adolescents is a growing and significant problem in Mexico. Given the high mortality rate associated with AIDS, the lack of available treatment, and the social stigma associated with the disease, prevention is the key to reducing the threat of AIDS among this important subgroup in Mexico. The study has four specific aims including 1) to determine whether the HIV risk-reduction intervention causes a greater increase in adolescents' intentions to abstain from intercourse and/or avoid unprotected intercourse at post-intervention and decreased self-reported intercourse and unprotected intercourse at 3, 6, 12, and 48 month follow-ups, compared with the general health promotion control intervention; 2) to determine whether the effects of the intervention are moderated by individual, microsystem, and macrosystem variables; 3) to identify theory-based variables that mediate effects of the HIV intervention on adolescents' self-reported behavior; and 4) to determine whether the HIV risk-reduction intervention causes a greater increase in parents' comfort with, and quantity of communication (general and HIV specific) with adolescents at post-intervention, 3, 6, 12, and 48 month follow-up compared with the general health promotion control intervention.

ELIGIBILITY:
Inclusion Criteria:

* Families (adolescents [aged 14 to 17 years of age] and one of their parents)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1620 (Actual)
Dates: Start 2002-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
General Parent-Adolescent Communication | pretest, posttest, 6 month follow-up, 12 month follow-up
Parent-Adolescent Sexual Risk Communication | Pretest, Posttest, 6 month follow-up, 12 month follow-up
Comfort With Communication | Pretest, Posttest, 6 month follow-up, 12 month follow-up
Intentions To Have Sexual Intercourse | Pretest, Posttest, 6 month follow-up, 12 month follow-up
  Questions regarding this measure were asked to adolescent participants only
Intentions to Use Condoms and Contraceptives | Pretest, Posttest, 6 month follow-up, 12 month follow-up
  Questions regarding this measure were asked to adolescent participants only

CONTACTS AND LOCATIONS:
Overall Officials: Antonia M. Villarruel, PhD, FAAN, Principal Investigator — University of Michigan
Locations (1):
- Preparatory Schools, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Result] Villarruel AM, Cherry CL, Cabriales EG, Ronis DL, Zhou Y. A parent-adolescent intervention to increase sexual risk communication: results of a randomized controlled trial. AIDS Educ Prev. 2008 Oct;20(5):371-83. doi: 10.1521/aeap.2008.20.5.371. PMID 18956979
- [Result] Gallegos EC, Villarruel AM, Loveland-Cherry C, Ronis DL, Yan Zhou M. [Intervention to reduce adolescents sexual risk behaviors: a randomized controlled trial]. Salud Publica Mex. 2008 Jan-Feb;50(1):59-66. doi: 10.1590/s0036-36342008000100012. Spanish. PMID 18297183
- [Result] Gallegos EC, Villarruel AM, Gomez MV, Onofre DJ, Zhou Y. Research brief: sexual communication and knowledge among Mexican parents and their adolescent children. J Assoc Nurses AIDS Care. 2007 Mar-Apr;18(2):28-34. doi: 10.1016/j.jana.2007.01.007. PMID 17403494
- See also: Curriculum materials (designed for Latino youth), overview of the curriculum, goals of the curriculum, types of activities, format and length, module outline, recommended training — http://www.selectmedia.org/customer-service/evidence-based-curricula/cuidate/